CLINICAL TRIAL: NCT05725148
Title: Prospective, Single-center, Single Group, Pivotal Clinical Trial to Evaluate the Blood Pressure Accuracy of 'CART-I Plus' Compared to the Reference Blood Pressure Reading With an Auscultatory Sphygmomanometer
Brief Title: Pivotal Clinical Trial to Evaluate the Blood Pressure Accuracy of 'CART-I Plus'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sky Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SL-BP-01
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Blood Pressure; Hypertension; Hypotension
Keywords: blood pressure
MeSH Terms: conditions — Hypertension; Hypotension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants whose SBP and DBP meet the ISO 81060-2:2018 requirements (Experimental): Each set of blood pressure tests is performed simultaneously. A cuff is worn on the right (or left) arm to check the blood pressure by auscultation, while 'CART-I plus' is worn on the finger of the opposite arm to check the blood pressure. At this time, the blood pressure test using an auscultation method is performed by two investigators simultaneously, and the blood pressure test using 'CART-I plus' is performed by the participants themselves
  Interventions: Device: CART-I plus

INTERVENTIONS:
Device: CART-I plus — CART-I plus is a ring-type medical device that continuously monitors Atrial Fibrillation, heart rate, oxygen saturation, and blood pressure using PPG and ECG signals.

SUMMARY:
The goal of this clinical trial is to evaluate how accurately the CART-I plus developed by Sky Labs can measure blood pressure. The primary endpoint of this clinical trial is accuracy (mmHg) of 'CART-I plus' which is obtained by calculating mean error and standard deviation of blood pressure differences between 'CART-I plus' and the gold standard for non-invasive method, auscultatory method. The reference readings are taken by auscultatory method using a sphygmomanometer and a stethoscope. The mean errors and standard deviations are calculated both sample- and subject-wise.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), hypertension is one of the major risk factors for death worldwide. The global adult population with hypertension is approximately 113 million, with an estimated prevalence of 18-27%. Hypertension is associated with stroke and other cardiovascular diseases, thus early detection and treatment critical. National guidelines of the Japanese, European, and American Hypertension Society recommend that home blood pressure and clinic blood pressure test results be applied together when diagnosing hypertension, emphasizing the importance of blood pressure monitoring in daily life. In addition, according to the Ohasama cohort study and the Finn-Home study, blood pressure measured in daily life was more predictive of cardiovascular disease than the office blood pressure.

There are invasive and non-invasive methods for blood pressure monitoring. The invasive method measures blood pressure using a pressure sensor by inserting a catheter into a blood vessel, and the non-invasive method measures blood pressure by sensing sound or vibration while applying pressure using a cuff. Invasive blood pressure tests can continuously measure blood pressure and are accurate, but there is a high risk of side effects such as distal ischemia, bleeding, thrombosis, infection, etc and is not available for a daily life. Non-invasive blood pressure test methods such as auscultatory measurement and oscillometric method are simpler than invasive methods, but it has limitations in measuring blood pressure continuously and observing long-term variations.

The photoplethysmography (PPG) method makes it possible to measure blood pressure without a cuff, enabling people to check and monitor blood pressure in daily life for a long time. It has been reported that the wavelength and amplitude of the PDW signal collected from the finger show a high correlation (0.92) with the PDP signal collected from the wrist. This suggests that the blood pressure accuracy of measuring blood pressure with PPG signals collected from the finger will not differ significantly from that measured from the wrist.

Sky Labs has developed 'CART-I plus' that can measure blood pressure in daily life without a cuff. 'CART-I plus' is a ring-type device that applies the principle of PPG technology to measure blood flow through finger veins. This clinical trial was designed in accordance with the ISO 81060-2:2018 standard to evaluate the accuracy of blood pressure estimated by 'CART-I plus'.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 19 or older
* Those who voluntarily decided to participate in this clinical trial and gave written consent to the subject explanation and consent form
* Those who is willing to comply with the clinical trial protocol

Exclusion Criteria:

* Those whose sound of fifth Kortkoff phase (K5) is not heard during blood pressure test using an auscultation type sphygmomanometer
* Those with unstable cardiac condition (myocardial infarction, ventricular arrhythmia, atrial fibrillation, premature ventricular contraction, pulmonary embolism 1 week before screening date)
* Those with arm circumference greater than 42 cm (> 42 cm)
* Those with a history of hypersensitivity to clinical trial medical device raw materials (PolyCarbonate, polycarbonate)
* Those with physical restrictions on wearing medical devices for clinical trials (for example, when ring-type clinical trial medical devices cannot be applied due to lack of appropriate ring size or other physical defects)
* Those who are judged to have difficulty collecting normal signals when wearing CART-I plus on a finger other than the thumb and forefinger (for example, if there is no CART-I plus model that fits the subject's finger)
* Those who is pregnant
* Those who is currently participating in other clinical trials or who have participated in other clinical trials within 30 days of the screening date
* Other cases where the investigator judges that participation in the clinical trial is inappropriate due to ethical reasons or may affect the results of the clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Accuracy of CART-I plus | 1 day
  Mean error and standard deviation of blood pressure differences between CART-I plus and reference (auscultatory method) readings

CONTACTS AND LOCATIONS:
Overall Officials: Seung Woo Park, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Sky Labs, Gyeonggi-do, Pangyo, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
The investigators would probably share the results showing the level of agreement between the two measurement methods after deidentification of participant data

REFERENCES:
- [Background] Ruiz-Rodriguez JC, Ruiz-Sanmartin A, Ribas V, Caballero J, Garcia-Roche A, Riera J, Nuvials X, de Nadal M, de Sola-Morales O, Serra J, Rello J. Innovative continuous non-invasive cuffless blood pressure monitoring based on photoplethysmography technology. Intensive Care Med. 2013 Sep;39(9):1618-25. doi: 10.1007/s00134-013-2964-2. Epub 2013 Jun 6. PMID 23740275
- [Background] Nachman D, Gepner Y, Goldstein N, Kabakov E, Ishay AB, Littman R, Azmon Y, Jaffe E, Eisenkraft A. Comparing blood pressure measurements between a photoplethysmography-based and a standard cuff-based manometry device. Sci Rep. 2020 Sep 30;10(1):16116. doi: 10.1038/s41598-020-73172-3. PMID 32999400
- [Background] Schoettker P, Degott J, Hofmann G, Proenca M, Bonnier G, Lemkaddem A, Lemay M, Schorer R, Christen U, Knebel JF, Wuerzner A, Burnier M, Wuerzner G. Blood pressure measurements with the OptiBP smartphone app validated against reference auscultatory measurements. Sci Rep. 2020 Oct 20;10(1):17827. doi: 10.1038/s41598-020-74955-4. PMID 33082436
- [Background] Watanabe N, Bando YK, Kawachi T, Yamakita H, Futatsuyama K, Honda Y, Yasui H, Nishimura K, Kamihara T, Okumura T, Ishii H, Kondo T, Murohara T. Development and Validation of a Novel Cuff-Less Blood Pressure Monitoring Device. JACC Basic Transl Sci. 2017 Dec 25;2(6):631-642. doi: 10.1016/j.jacbts.2017.07.015. eCollection 2017 Dec. PMID 30062178
- [Background] Pellaton C, Vybornova A, Fallet S, Marques L, Grossenbacher O, De Marco B, Chapuis V, Bertschi M, Alpert BS, Sola J. Accuracy testing of a new optical device for noninvasive estimation of systolic and diastolic blood pressure compared to intra-arterial measurements. Blood Press Monit. 2020 Apr;25(2):105-109. doi: 10.1097/MBP.0000000000000421. PMID 31688003
- [Background] Stergiou GS, Alpert B, Mieke S, Asmar R, Atkins N, Eckert S, Frick G, Friedman B, Grassl T, Ichikawa T, Ioannidis JP, Lacy P, McManus R, Murray A, Myers M, Palatini P, Parati G, Quinn D, Sarkis J, Shennan A, Usuda T, Wang J, Wu CO, O'Brien E. A Universal Standard for the Validation of Blood Pressure Measuring Devices: Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO) Collaboration Statement. Hypertension. 2018 Mar;71(3):368-374. doi: 10.1161/HYPERTENSIONAHA.117.10237. Epub 2018 Jan 31. PMID 29386350
- [Background] Tsai PY, Huang CH, Guo JW, Li YC, Wu AA, Lin HJ, Wang TD. Coherence between Decomposed Components of Wrist and Finger PPG Signals by Imputing Missing Features and Resolving Ambiguous Features. Sensors (Basel). 2021 Jun 24;21(13):4315. doi: 10.3390/s21134315. PMID 34202597